CLINICAL TRIAL: NCT02548065
Title: Efficacy and Tolerability of Balneotherapy With Mineral Water Named" Debole of Vetriolo" in Patients With Fibromyalgia Syndrome (FS): A Randomized Double Blind Controlled Clinical Trial
Brief Title: Efficacy and Tolerability of Balneotherapy With Mineral Water Named" Debole of Vetriolo" in Fibromyalgia Syndrome
Acronym: VET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Senese (Other)
Responsible Party: Principal Investigator, Fioravanti Antonella, Assistant of Professor, Azienda Ospedaliera Universitaria Senese
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AOUSenese
Record Dates: First submitted 2015-09-04; First posted 2015-09-14 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Fibromyalgia Syndrome
Keywords: Fibromyalgia Syndrome; Balneotherapy; Vetriolo Water
MeSH Terms: conditions — Fibromyalgia | interventions — Balneology

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Balneotherapy (Active Comparator): Daily thermal-mineral bath with mineral water named "Debole of Vetriolo" for a total of 12 applications carried out over a period of two weeks at Levico Terme Spa Center (Levico Terme, Italy)
  Interventions: Other: Balneotherapy
- Placebo (Placebo Comparator): daily thermal bath with tap water bath for a total of 12 applications carried out over a period of two weeks at Levico Terme Spa Center (Levico Terme, Italy)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Balneotherapy — Bath with mineral water named "Debole of Vetriolo" at 36°C, 15 minutes for 12 consecutive days in bathtubs
  Other Names: spa therapy
  Arms: Balneotherapy
Other: Placebo — Bath with Thermal tap water
  Other Names: Tap water
  Arms: Placebo

SUMMARY:
The present randomized, controlled double blind trial aims to evaluate the efficacy and tolerability of balneotherapy with mineral water named "Debole of Vetriolo" in 100 patients with primary Fibromyalgia Syndrome (FS).

DETAILED DESCRIPTION:
The fibromyalgia syndrome (FS) is a chronic condition that is characterized by chronic widespread pain, fatigue, sleep disorders, cognitive disturbances, physical and psychological distress. It was estimated that between 2.9 and 3.8% of the general population in Europe and the US are affected , with the majority of patients in clinical settings being female . Clinical research suggests that pharmacologic treatment alone is not the best approach for FS, and that an integrated approach that includes non-pharmacologic therapies along with pharmacologic therapies improves outcomes in these patients.

Balneotherapy is one of the most commonly used non-pharmacological approaches for SF, but it is still being discussed and its role in modern medicine is still not clear. The action mechanisms of thermal baths are not completely known, and it is difficult to distinguish the effects of thermal applications from the benefits that could be derived from a stay in a spa environment.

The present randomized, controlled double blind trial aims to evaluate the efficacy and tolerability of balneotherapy with mineral water named "Debole of Vetriolo" in patients with primary SF fulfilling the 2010 ACR criteria.

Following confirmation that the patients fulfill the screening criteria and having obtained written informed consent, 100 patients will be randomized 1:1 and allocated to one of two groups using a computer-generated table of random numbers:

Group I (50 patients) will be treated with daily thermal-mineral bath with mineral water named "Debole of Vetriolo" for a total of 12 applications carried out over a period of two weeks at Levico Terme Spa Center (Levico Terme, Italy)

Group II (50 patients), the control group, will be treated with daily thermal bath with with tap water bath for a total of 12 applications carried out over a period of two weeks at Levico Terme Spa Center (Levico Terme, Italy)

The block randomization list will be kept by individuals who have no contact with the investigators who assign patients to their randomized treatment, and who will not perform any patient assessment or conduct the statistical.

All patients will undergo general medical evaluation and rheumatologic examination by the same physician before the start of the study. All the demographic, anamnestic and clinical data will be collected on identical questionnaires. Each patient will be assessed at baseline time (T0), after 2 weeks (T1),after 3 months (T2), 6 months (T3), following the beginning of the study.

All assessments will be performed at Levico Terme Spa Centre by the same rheumatologist who will be blinded to which study arms the patients belongs. Laboratory analysis will be performed only at baseline.

Assessments at each examination will include:

Primary Outcome Measures

* Visual Analogue Scale (VAS);
* Fibromyalgia Impact Questionnaire total score (FIQ-Total) e Fibromyalgia Impact Questionnaire Physical score (FIQ-PI)

Secondary Outcome Measures

* Widespread Pain Index (WPI)
* Symptom Severity (SS)
* Short Form Health Survey (SF-12)
* State-Trait Anxiety Inventory (STAI)
* Center for Epidemiologic Studies Depression Scale (CES-D)

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from FS according to American College of Rheumatology (ACR) criteria for at least 3 months and with a stable treatment for at least 4 weeks
* Have a score of WPI≥7 and SS ≥ 5 or WPI 3-6 and SS≥9 screening and baseline visit
* Provide written informed consent to participate in the study

Exclusion Criteria:• Concurrent participation in other therapeutic trials

* Patients that have been treated with mud-pack therapy and/or balneotherapy in the last 6 months
* Patients affected by neoplastic diseases in the last five years, with cardiovascular disease of recent onset, suffering from serious impairment of hematopoietic, renal and hepatic systems
* Presence of concurrent autoimmune or inflammatory disease, such as, rheumatoid arthritis, systemic lupus erythematous, inflammatory bowel disease, etc.
* Pregnant and nursing mothers
* Severe psychiatric illnesses (current schizophrenia, major depression with suicidal ideation, within two years)
* Routine daily use of narcotic analgesics or history of substance abuse
* Patients unable to complete the questionnaires

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
Change of 20% of VAS score | change from baseline at 15 days
  VAS score,
Change of 20% Total FIQ | change from baseline at 15 days
  FIQ

SECONDARY OUTCOMES:
Quality of life assessed by SF-12 | Baseline time , after 2 weeks ,after 3 months, 6 months, following the beginning of the study.
  SF-12
Anxiety evaluation by STAI | Baseline time , after 2 weeks ,after 3 months, 6 months, following the beginning of the study.
  STAI
Depression assessed by CES-D | Baseline time , after 2 weeks ,after 3 months, 6 months, following the beginning of the study.
  CES-D
Widespread Pain assessed by WPI | Baseline time , after 2 weeks ,after 3 months, 6 months, following the beginning of the study.
  WPI
Symptom Severity assessed by SS scale | Baseline time , after 2 weeks ,after 3 months, 6 months, following the beginning of the study.
  SS

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Fioravanti, MD, Principal Investigator — Azienda Ospedaliera Universitaria Senese
Locations (1):
- Fioravanti Antonella, Siena, Siena, Italy

REFERENCES:
- [Background] Guidelli GM, Tenti S, De Nobili E, Fioravanti A. Fibromyalgia syndrome and spa therapy: myth or reality? Clin Med Insights Arthritis Musculoskelet Disord. 2012;5:19-26. doi: 10.4137/CMAMD.S8797. Epub 2012 Feb 22. PMID 22408369
- [Background] Buskila D, Abu-Shakra M, Neumann L, Odes L, Shneider E, Flusser D, Sukenik S. Balneotherapy for fibromyalgia at the Dead Sea. Rheumatol Int. 2001 Apr;20(3):105-8. doi: 10.1007/s002960000085. PMID 11354556
- [Background] Neumann L, Sukenik S, Bolotin A, Abu-Shakra M, Amir M, Flusser D, Buskila D. The effect of balneotherapy at the Dead Sea on the quality of life of patients with fibromyalgia syndrome. Clin Rheumatol. 2001;20(1):15-9. doi: 10.1007/s100670170097. PMID 11254234
- [Background] Evcik D, Kizilay B, Gokcen E. The effects of balneotherapy on fibromyalgia patients. Rheumatol Int. 2002 Jun;22(2):56-9. doi: 10.1007/s00296-002-0189-8. Epub 2002 Mar 29. PMID 12070676
- [Background] Donmez A, Karagulle MZ, Tercan N, Dinler M, Issever H, Karagulle M, Turan M. SPA therapy in fibromyalgia: a randomised controlled clinic study. Rheumatol Int. 2005 Dec;26(2):168-72. doi: 10.1007/s00296-005-0623-9. Epub 2005 Jun 17. PMID 15965635
- [Background] Fioravanti A, Perpignano G, Tirri G, Cardinale G, Gianniti C, Lanza CE, Loi A, Tirri E, Sfriso P, Cozzi F. Effects of mud-bath treatment on fibromyalgia patients: a randomized clinical trial. Rheumatol Int. 2007 Oct;27(12):1157-61. doi: 10.1007/s00296-007-0358-x. Epub 2007 May 23. PMID 17520260
- [Result] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783
- [Derived] Fioravanti A, Manica P, Bortolotti R, Cevenini G, Tenti S, Paolazzi G. Is balneotherapy effective for fibromyalgia? Results from a 6-month double-blind randomized clinical trial. Clin Rheumatol. 2018 Aug;37(8):2203-2212. doi: 10.1007/s10067-018-4117-z. Epub 2018 May 5. PMID 29730741